CLINICAL TRIAL: NCT06864364
Title: Effect of Continuous Glucose Monitoring on Perceived Benefits of a Milk With Mulberry Leave Extract in Non-diabetic Adult Chinese Population
Brief Title: Effect of Visualization of Functional Milk Efficacy on Perceived Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2301NR
Record Dates: First submitted 2025-02-06; First posted 2025-03-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy; Prediabetes; Asian; Adult
Keywords: CGM; perceived benefit
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visualization (intervention arm, group A) (Experimental): CGM feedback visualization
  Interventions: Other: CGM feedback visualization; Dietary Supplement: milk supplemented with mulberry leaves extract
- Blinded Visualization (control arm, group B) (Placebo Comparator): blinded for CGM feedback visualization
  Interventions: Dietary Supplement: milk supplemented with mulberry leaves extract; Other: blinded CGM feedback visualization

INTERVENTIONS:
Other: CGM feedback visualization — The subject will have CGM feedback visualization
  Arms: Visualization (intervention arm, group A)
Dietary Supplement: milk supplemented with mulberry leaves extract — milk supplemented with mulberry leaves extract
Other: blinded CGM feedback visualization — The subject will have blinded CGM feedback visualization
  Arms: Blinded Visualization (control arm, group B)

SUMMARY:
This study aims to demonstrate the effect of visualizing the effect of consuming a functional milk on postprandial glucose response on perceived benefits compared to absence of visualization.

DETAILED DESCRIPTION:
This is a multi-centric double-blind, randomized, 2-arm parallel group clinical study to investigate the effect of of consuming a functional milk on postprandial glucose response on perceived benefits compared to absence of visualization.

The study is divided in 3 periods: 1) reference period in which both groups will have a blinded Continuous Glucose Monitoring (CGM) sensor; 2) intervention period where participants will have either CGM feedback visualization or blinded CGM feedback visualization, while both arms consume a functional milk powder; 3) follow-up in free-living conditions.

Outcomes of this study will include plasma HbA1c, glucose, insulin and lipids levels, perceived benefits and adherence questionnaire, dietary intake and physical activity and real usage.

This will be conducted in a total of 170 healthy adults of Chinese ethnicity aged 45-75 years

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand and sign a written informed consent prior to study entry
2. Deemed able to comply with the requirements of the study protocol and consume study product
3. BMI: 18.5-35.0 kg/m2 (inclusive)
4. Age: 45-75y (inclusive 45 and 75)
5. Males and females
6. HbA1c ≤ 6.4 % and FPG ≤ 6.90 mmol/L (125 mg/dl) to exclude diabetic individuals based on the National Institute of Health and Care (NICE) criteria
7. Regularly consuming a carbohydrate containing breakfast (≥30g of total CHO) assessed by a food recall only at breakfast of the previous day to the screening visit
8. Having a sedentary lifestyle meaning do not usually conduct vigorous*-intense physical activity and are willing to abstain from it during reference and intervention period
9. If on chronic medication such as lipid-lowering, thyroid medication, etc., the dosage must be constant for at least 3 months prior to screening.

   * Activities such as jogging, running, carrying heavy objects or other loads upstairs, shoveling snow, participating in a fitness class, and fast swimming, that will lead to hard and fast breathing.

Exclusion Criteria:

1. Pre-existing chronic medical condition and/or history of significant medical condition (e.g. malignancy, significant organ dysfunction, autoimmune and/ or genetic disease, gastrointestinal disease, endocrine disease (e.g. diabetes mellitus, history of hypoglycemia, polycystic disease syndrome, Addison's disease, Cushing's syndrome, acromegaly), acute or chronic infectious condition (e.g. hepatitis B and C, HIV, tuberculosis), cardiovascular disease (heart failure, angina, myocardial infarction, stroke), renal disease (renal insufficiency), hepatic (liver cirrhosis, liver failure) or respiratory disease (COPD), hematological disorder (e.g. anemia), neurological and/or psychiatric conditions (e.g. depression, psychotic disorders, chronic insomnia eating disorder), as diagnosed by the treating physician, which in the opinion of the site physician/ investigator may risk participant wellbeing/ safety, impede participant compliance with study procedures or ability to complete the study and/ or could confound the primary objectives of the study.
2. Any acute illness or any recent medical/ surgical intervention within 3 months prior to enrolment potentially interfering with study procedures and assessments.
3. Known or suspected cow's milk protein allergy (CMPA), lactose and /or soy intolerance /hypersensitivity.
4. Known substance abuse or alcohol user exceeds following intake on a regular basis, alcohol intake > 2 servings per day for males and > 1 servings per day for females. A serving is 40ml of strong alcohol, 100 ml of red or white wine, or 300 ml of beer.
5. Current smoker (e.g., cigarette, tobacco, cannabis) who exceeds 5 cigarettes per week.
6. Patients with refractory hypertension, and patients with hypertension who are taking antihypertensive drugs (beta-blockers, thiazide diuretics) that may affect blood glucose metabolism.
7. Female participants currently on hormonal therapy including post-menopausal hormone Replacement Therapy (PRT) or have been on PRT treatment in the past two months before study participation.
8. Participants on systemic corticosteroids, glucocorticoids, or cyclosporine A.
9. Female participants who are pregnant or intending to become pregnant, lactating and or breastfeeding.
10. Participants who had a significant weight loss (≥5%) within the last 6 months or follow a weight loss programme.
11. Following diets with low carbohydrate content (e.g., ketogenic diet, Atkins diet, low-carb diet, carb cycling diet), intermittent fasting, breakfast skippers or any self-restricted, controlled, or special therapeutic diet.
12. Participants who do not regularly (≤ 3 times per week) drink dairy milk.
13. Use of multivitamin/ multimineral supplements (including vitamin C, supplements fiber-based or derived of leaf extracts or known to/intended to lower blood glucose as per package claim) up to 15 days prior to screening.
14. Medically known cutaneous hypersensitivity to adhesives, silicon watchstrap and plasters.
15. High daily coffee consumption (≥400 mg of caffeine/day, equivalent to ≥4 cups of coffee).
16. Currently participating in another interventional clinical study.
17. Having two (or more) participants from the same household already enrolled in the study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Likert-scale for perceived benefit | From enrollment to day 30
  A Likert-scale from 1 (very unlikely) to 7 (very likely) on perceived product benefits

SECONDARY OUTCOMES:
Likert-scale for product experience | From enrollment to day 15 and day 30
  A Likert-scale from 1 (very unlikely) to 7 (very likely) on product experience.
Likert-scale for perceived benefit | From enrollment to day 15
  A Likert-scale from 1 (very unlikely) to 7 (very likely) on perceived product benefits.
Actual usage and recommendation behavior | At day 88
  Actual usage and recommendation behavior will be measured comparing answers at the end of the follow up period (V6) from Group A vs. Group B to 5 questions generated for this study.
  1. Have you bought Yiyang TangLv since the intervention ended (visit 5)? Yes No 1.1 If so, how many tins or/and sachet did you buy? (Specify number) This includes for yourself or family ___ tins
     * sachets
  2. How often have you drank Yiyang TangLv since the end intervention (visit 5)? Never <3 times a week 4-6 days a week 7 days a week
  3. Did you drank it in the morning with breakfast? Yes No
  4. Has anyone else in your household drank Yiyang TangLv since the intervention ended (visit 5)? Yes No not sure
  5. Have you recommended Yiyang TangLv to anyone since the study end of the intervention (visit 5)? Yes No
CGM markers - iAUC0-60,120,180 min post-breakfast | From enrollment to day 30
  Changes in CGM markers in response to IP intake (mmol/L x min) .
CGM markers - 24h iAUC | From enrollment to day 30
  Changes in CGM markers. (mmol/L x min)
CGM markers - iCmax | From enrollment to day 30
  Changes in CGM markers in response to IP intake (mmol/L) .
CGM markers - Tmax | From enrollment to day 30
  Changes in CGM markers in response to IP intake (min).
CGM markers - time in range (TIR) | From enrollment to day 30
  Changes in CGM markers (%).
CGM markers - average interstitial glucose | From enrollment to day 30
  Changes in CGM markers (mmol/L).
CGM markers - coefficient of variance (CV) | From enrollment to day 30
  Changes in CGM markers (%) .
CGM markers - mean amplitude of glycaemic excursion (MAGE) | From enrollment to day 30
  Changes in CGM markers (mmol/L) .

OTHER OUTCOMES:
Long-term glucose metabolism -HbA1c | From day 0 to day 88
  HbA1c (%) changes
International physical activity questionnaire | From enrollment to day 88
  Changes in physical activity levels captured via the International physical activity questionnaire (IPAQ), category: low, moderate, high
Macronutrient and energy intake | From enrollment to day 88
  Changes in dietary intake measured using 3-day-food diaries
Actual changes in perceived change in lifestyle | From enrollment to day 88
  Actual changes in perceived change in lifestyle will be measured by answering questions:
  1 Do you feel that continuous glucose monitor use contributed to you making changes for a healthier lifestyle? (Yes/No/Not sure) 2. After continuous glucose monitor use, do you feel that you changed your diet by limiting or including certain foods? (Yes/No/Not sure) 3. Do you think continuous glucose monitor use made you more likely to be more active/increase your exercise? (Yes/No/Not sure)
App usage - App screen time | From enrollment to day 30
  Understanding of the app usage will be measured throughout the intervention period with metric of App screen time
Long-term glucose metabolism -fasting plasma glucose | From day 0 to day 88
  fasting plasma glucose (mmol/L) changes
Long-term glucose metabolism -insulin levels | From day 0 to day 88
  insulin levels ( μU/mL) changes
Long-term glucose metabolism -HOMA-IR | From day 0 to day 88
  HOMA-IR (numerical index) changes
lipid metabolism changes - HDL-C | From day 0 to day 88
  HDL-C (mmol/L) changes
lipid metabolism changes - LDL-C | From day 0 to day 88
  LDL-C(mmol/L)changes
lipid metabolism changes -Total cholesterol | From day 0 to day 88
  Total cholesterol (mmol/L) changes
lipid metabolism changes - Triglycerides | From day 0 to day 88
  Triglycerides(mmol/L)changes
Weight outcomes changes - waist circumference | From day 0 to day 88
  waist circumference(cm)changes
Weight outcomes changes - BMI | From day 0 to day 88
  weight and height will be combined to report BMI in kg/m^2 , and the changes of BMI.
Weight outcomes changes - Body weight, | From day 0 to day 88
  Body weight (kg) changes
App usage - numbers of log per days | From enrollment to day 30
  Understanding of the app usage will be measured throughout the intervention period with metric of number of log per days.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China